CLINICAL TRIAL: NCT05560113
Title: Forgetting Fear: Establishing a Novel Non-invasive Approach to Disrupt Fear-based Sensory Memory Consolidation in Humans
Brief Title: Disrupting Fear-based Memory Consolidation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael R Borich, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004510
Record Dates: First submitted 2022-09-15; First posted 2022-09-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Fear; Transcranial Magnetic Stimulation; Memory
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS: Inhibitory Transcranial magnetic stimulation (TMS) to sensory Cortex (Experimental): Participants will undergo a Functional magnetic resonance imaging (fMRI) scan while performing a fear conditioning/extinction task at the Center for Systems Imaging- Emory University Hospital (CSI-EUH) and then either stay at CSI-EUH or relocate to the Neural Plasticity Research Laboratory at Emory Rehabilitation Hospital. Participants will then be randomly assigned to either receive active or sham continuous theta burst stimulation (cTBS) to transiently disrupt neural activity in the targeted sensory cortex region specifically during the sensory memory consolidation window.
  Interventions: Other: Continuous theta burst stimulation (cTBS)
- Sham cTBS (Placebo Comparator): Participants will undergo a Functional magnetic resonance imaging (fMRI) scan while performing a fear conditioning/extinction task at CSI-EUH and then either stay at CSI-EUH or relocate to the Neural Plasticity Research Laboratory at Emory Rehabilitation Hospital. Participants will then be randomly assigned to either receive active or sham continuous theta burst stimulation (cTBS) to transiently disrupt neural activity in the targeted sensory cortex region specifically during the sensory memory consolidation window.
  Interventions: Other: Sham continuous theta burst stimulation (cTBS)

INTERVENTIONS:
Other: Continuous theta burst stimulation (cTBS) — cTBS, a patterned form of TMS, (80% active motor threshold intensity, 3 pulses at 50Hz, 200ms interval, 600 pulses, 40s duration applied over the targeted sensory cortical region using real-time neuronavigation to focally and transiently inhibit neural activity
  Arms: cTBS: Inhibitory Transcranial magnetic stimulation (TMS) to sensory Cortex
Other: Sham continuous theta burst stimulation (cTBS) — This will be a sham intervention. An active/sham stimulating coil will be used for double-blinding of stimulation condition. cTBS is safe and has established safety guidelines that will be strictly adhered to during study conduction.
  Arms: Sham cTBS

SUMMARY:
This project represents a unique collaborative opportunity to pursue the essential proof-of-principle demonstration that non-invasive interference of sensory cortical memory consolidation shortly after an emotional experience can attenuate the cued fear response and potentially reduce the risk of developing post-traumatic stress disorder (PTSD). If successful, the study results would anchor a potential advance in the treatment of patients after a traumatic event and seed future animal and clinical studies of emotional sensory cortical memory consolidation to reduce the prevalence and negative sequelae of PTSD.

DETAILED DESCRIPTION:
This mechanistic study in humans will study an unexplored precision-based approach of non-invasive neuromodulation of sensory cortex with the aim to prevent PTSD by attenuating the sensory encoding of fear memory. The objective of this project is to explore the basic science and therapeutic potential of sensory-emotional reprogramming in humans, and translate this idea into a precise, individualized treatment to reduce the risk that negative emotional sensory experiences lead to PTSD. Understanding sensory-emotional programming in humans could anchor a breakthrough in the treatment of patients after a traumatic event and seed future animal and clinical studies of emotional sensory cortical memory consolidation to reduce the prevalence and negative sequela of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Willingness to participate in study
* No history of musculoskeletal impairment or neurological disease
* Clinical diagnosis of PTSD for individuals in the PTSD group.

Exclusion Criteria:

* Any participant outside the age range
* Participants that show signs of dementia (score < 20 on the Montreal Cognitive Assessment)
* Participants that have a history of major head trauma, a neurodegenerative disorder, or recent (<6 months) substance abuse;
* Participants that had a recent history of Central Nervous System (CNS) active drugs that may influence cortical excitability or learning; or
* Participants that report contraindications to TMS or MRI - if participating in the TMS/MRI experiments
* Current psychoactive medication usage
* Current symptoms of psychosis or bipolar disorder (as indicated by study staff through a clinical interview as part of that study).
* The study will exclude adults unable to consent, individuals who are not yet adults, pregnant women and prisoners on scientific grounds and to minimize risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Neural Connections: Functional network connectivity | Study Day 30 and Day 31
  Preprocessing of neuroimaging data will be conducted using fMRI prep. Pre-processed neuroimaging data will undergo first and second level modeling in Statistical Parametric Mapping. First level analysis include an event-related model with the onset and duration of each event included for each condition, and motion included as a regressor. A high-pass filter of 128s will be applied to account for low-frequency drifts. Amygdala regions of interest (ROIs) will be defined anatomically using California Institute of Technology (CIT168) Subcortical Atlas. Primary sensory cortex ROI & seed coordinates will be defined utilizing voxels within a V1 region mask showing maximal functional connectivity with the amygdala during conditioning.
Changes in Neural Connections: Regional activation | Study Day 30 and 31
  Preprocessing of neuroimaging data will be conducted using fMRI prep. Pre-processed neuroimaging data will undergo first and second level modeling in Statistical Parametric Mapping. First level analysis include an event-related model with the onset and duration of each event included for each condition, and motion included as a regressor. A high-pass filter of 128s will be applied to account for low-frequency drifts. Whole-brain analysis of changes in local regions of activity will be measured by change in blood-oxygen-level-dependent (BOLD) signal from resting activity. Multiple comparisons using permutation-based methods to control the false positive rate to p<.05.

SECONDARY OUTCOMES:
Changes in Measures of skin conductive response | Study Day 30 and Day 31
  Skin conductance response (SCR) will be recorded during localization, conditioning, and fear retention tasks using the BIOPAC system MP150 (BIOPAC systems, Inc.) and parameters previously utilized in the lab. SCR is a validated physiological measure of sympathetic arousal, with higher SCR indicating a higher arousal response to conditioned stimuli. Change in SCR from early to late extinction is our primary indicator of the degree of extinction learning. SCR will be scored as a response to individual Conditioned Stimulus (CS)+E and CS- stimuli (maximum SC within 6 seconds post-CS onset, minus average SC over a 2-second prestimulus baseline) and will be square-root transformed for normalization. Early fear extinction will be defined as occurring within the first fear extinction run, with late fear extinction being defined as the second extinction run.
ECG | Study Day 31
  Heart rate and heart-rate variability (HRV) will be measured using the ECG module of the BIOPAC system at a sampling rate of 1 kilo Hertz (kHz). One 5mm Ag/AgCl (Silver/Silver Chloride) electrode will be placed on the chest above the right clavicle, another electrode will be placed on the chest under the left side of the ribcage.
Acoustic Startle response | Study Day 31
  The acoustic startle response (eyeblink component) will be measured via electriomyography (EMG) of the right orbicularis oculi muscle. Two 5 mm Ag/AgCl pre-gelled disposable electrodes will be positioned approximately 1 cm under the pupil and 1 cm below the lateral canthus. The startle probe (noise burst) will be a 108-decibel (dB) (A) Sound Pressure Level (SPL), 40-ms burst of broadband noise with a near instantaneous rise time . The startle probe is a white noise burst that is affectively neutral and clearly differentiable from the aversive sound used for the US.
Changes in Fear conditioning and extinction task | Study Day 30 and Day 31
  Participants will view pictures of animals and tools which will not be repeated. During the 1st phase, 3 categories of images will be displayed: animals, tools, and animal/tool images phase-scrambled. Blocks of 10 images of each category will be displayed 4 times, with each image displayed for 0.75 seconds with a 0.25 s delay between images and 11 s inter-block interval. This task will allow for localization of brain areas activated by animal images vs. tool images, with the phase scrambled images serving as a control. 15 animal and 15 tool images will be randomly displayed for 4.5 s with a fixation cross displayed between each image for 6, 8, or 10 seconds. For the 2nd phase, 10 of either the animal or tool images are assigned as the CS+, and paired with the US, a 1-second loud screeching sound at the end of the image presentation. The other image type, the CS-, will not be paired with the US. In the fear retention phase on Day 2, the CS+ and CS- will be presented without the US.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borich, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Rehabilitation Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Raw and preprocessed magnetic resonance imaging data as well as behavioral data.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available after completion of primary data analyses.
Access Criteria: : Data will be made publicly available using a data archive (e.g., IPD Sharing Statement LONI Laboratory of Neuro Imaging (LONI), ida.loni.usc.edu) for potential big data analyses as well as reproducibility analyses